CLINICAL TRIAL: NCT03999450
Title: Preventing Premature Death Among Hospital Patients With Serious Opioid-Related Infection (SORI): A Phase 1 Pilot Study
Brief Title: Preventing Premature Death in Patients With Serious Opioid-related Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Marc Swogger, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RSRB00003696
Record Dates: First submitted 2019-06-05; First posted 2019-06-26 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Opioid Use
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral intervention (Experimental): Patients admitted to Strong Hospital with opioid use will be given 1 to 3 brief motivational interventions and computer based cognitive behavioral therapy
  Interventions: Behavioral: brief motivational intervention (BMI); Behavioral: cognitive behavioral therapy

INTERVENTIONS:
Behavioral: brief motivational intervention (BMI) — The intervention typically takes 45 minutes to administer and is designed to enhance motivation to change and includes the following components: establishing rapport, asking permission to discuss substance use and providing feedback regarding the substance use assessment, exploring personal consequences of drug use, eliciting the gap between real and desired quality of life, and discussing readiness to change. The therapist then negotiates a written action plan, during which the subject is supported with empathy and verbal reinforcement.
Behavioral: cognitive behavioral therapy — This evidence-based, online, Computer Based Training for Cognitive Behavioral Therapy (CBT4CBT) program covers six lessons: 1) changing patterns of use, 2) coping with craving, 3) refusing drugs, 4) problem-solving skills, 5) changing drug-related thoughts, and 6) improving decision-making. The program is designed to be user-friendly and includes videotaped instructions and examples, interactive assessments, and practice exercises.

SUMMARY:
The purpose of this study is to test the efficacy of a combination of motivational interventions and a brief therapy session to increase the adherence to medication-assisted treatment (MAT) for opioids.

DETAILED DESCRIPTION:
We will recruit 30 SORI inpatients ages 18-plus admitted to the University of Rochester Medical Center (URMC). We will administer a battery of validated assessments of substance use, overdose history and risk, opioid-related infection, and suicidal behavior at baseline and approximately 2- and 4-week follow-ups. We will assess both forms of overdose (unintentional, intentional - i.e., suicidal behavior) because each is common in intravenous drug users and they require systematic assessment to disentangle. All recruited individuals will receive one-to-three MI sessions as they begin the MAT that is part of standard hospital care. Patients will be offered computer-based CBT, which they will complete on the unit at their convenience. The CBT program records duration of use of the treatment modules, enabling us to track patients' level of CBT treatment participation. Patient-completed intervention feedback forms and treatment completion will be examined after 15 subjects have participated. Based on this feedback, we will pilot an adapted (MI plus CBT) treatment manual, obtaining additional feedback on acceptability. We will assess psychopathy, a constellation of stable traits and potentially important moderator of treatment effects, at baseline. We will assess potential mediators (i.e., motivation to change, self-regulation) using validated measures at baseline and at approximately 2- and 4-weeks post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide contact information (e.g., email, phone, address)
* Presence of SORI, including endocarditis, osteomyelitis, septic arthritis, epidural abscess, or serious bacteremia
* Hospital length of stay estimated at > 3 weeks
* Admitted to URMC and seen by the Toxicology Consult Team. Providers will be informed of inclusion/exclusion requirements so that they can make an informed decision about whether a patient may be approached.

Exclusion Criteria:

* Non-English speaking
* Unwilling to provide informed consent; unable to provide informed consent or participate in study procedures due to lack of comprehension, medical barriers (e.g., intubated), or behavioral (e.g., violence) or severe psychiatric problems (e.g., florid psychosis). Capacity to provide informed consent will be determined by their treatment team or other provider consult team as appropriate. This serves a dual function of both basing consent capacity on the most accurate and current medical information, as well as keeping their treatment team informed of any research involvement of their patient.
* Note that patients may be ineligible initially but become eligible due to stabilization during hospitalization, at which point we would then proceed as usual with the identification and recruitment process. We will seek to recruit every SORI admission who meets eligibility criteria within the recruitment timeframe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who completed the week 4 follow up assessments | week 4
  The percentage of participants who completed the week 4 follow up assessments.
Percentage of participants who report intervention acceptability | week 4
  Written and verbal feedback will be collected from participants.
Change in mean readiness | baseline to 2 weeks
  A readiness ruler with a scale of 1- 10 where higher numbers indicate better health outcomes will be used to to assess motivation to change illicit substance use.
Change in mean self-regulation | baseline to 2 weeks
  The Self-Regulation Questionnaire is a 63 item questionnaire with each question rated at a 5-point likert scale.
  > 239 High (intact) self-regulation capacity (top quartile) 214-238 Intermediate (moderate) self-regulation capacity (middle quartiles) < 213 Low (impaired) self-regulation capacity (bottom quartile)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided